CLINICAL TRIAL: NCT06191484
Title: Risk and Resilience to Late-life Suicidal Ideation and Behavior After Spousal Bereavement: Targeting Social Connectedness to Strengthen Circadian Rhythmicity
Brief Title: Risk and Resilience to Suicide Following Late-Life Spousal Bereavement
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah T. Stahl, PhD, Associate Professor of Psychiatry and Assistant Professor of Clinical and Translational Science, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY23060037; R01MH132114 (NIH)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Suicide; Bereavement
Keywords: grief; bereavement; suicide; geriatric; health; technology; depression
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WELL Behavioral Probe (Experimental): Digital monitoring of sleep, meals, and social activity, for 3 months.
  Interventions: Behavioral: WELL Behavioral Probe

INTERVENTIONS:
Behavioral: WELL Behavioral Probe — Participant record the timing and regularity of sleep, meals, and social activity twice daily, for 3 months, using a digital diary. Participants also receive weekly motivational health coaching.

SUMMARY:
The purpose of the RISE study is to examine how the 24-hour rhythm of sleep and social activity relate to mood and suicidal ideation among older adults that recently lost a spouse or life partner.

DETAILED DESCRIPTION:
Experiencing the death of a spouse or life partner is a profoundly distressing event that may cause abrupt changes in one's daily routine, including decreased self-care and withdrawal from social activities. While most individuals adapt over time, a substantial number of older bereaved spouses (20-35%) experience depression, loneliness, suicidal thoughts, and early mortality, including death by suicide.

The objective of this study is to examine the risk for and resilience to late life suicide during the early spousal bereavement period by investigating the extent to which (1) social connectedness influences suicide risk and (2) whether circadian rhythm instability (inconsistent patterns of sleep, activity, meals, and socialization) helps explain this association.

The investigators will enroll 169 adults aged 60+ years who experienced the death of a spouse or life partner within the previous 12 months. All participants will complete repeated assessments of social connectedness, clinical assessments of depression and suicide ideation, and accelerometry recordings of the 24-hour pattern of sleep and activity. Participants will also complete a 3-month behavioral probe, designed to promote self-care behaviors in older bereaved spouses using technology and motivational health coaching. The behavioral probe targets circadian rhythm stability by focusing on regular routine of sleep, meals, and social activities. The behavioral probe will determine whether modifying social connectedness reduces suicide risk and whether circadian rhythm stability explains part of this association.

ELIGIBILITY:
Older adults who recently lost their spouse or life partner and are high risk for suicidal thoughts and/or behavior.

Inclusion Criteria:

1. Bereaved < or = to 12 months from spousal/partner loss
2. > or = to 65 years old
3. Verified history of suicide attempt/attempts and/or current or past history of Major Depressive Disorder/Major Depressive Episode (MDD/MDE) (without psychotic features), or history of depression severe enough to trigger treatment, or current subsyndromal depression (> or = to 9 HDRS)
4. No diagnosis of schizophrenia/schizoaffective disorders/bipolar/current psychosis
5. Does not reside in nursing home
6. Not a current shift worker
7. No major cognitive impairment: TICS score of > or = to 27

Exclusion Criteria:

1. Bereaved >12 months from spousal/partner bereavement
2. < 65 years old
3. Patient is not spousal/partner bereaved (ex: parent, sibling, etc.)
4. Prior diagnosis of schizophrenia/schizoaffective disorders/bipolar/current psychosis or medications listed indicate diagnosis of these disorders/MDD or MDE with psychotic features
5. Major cognitive impairment: TICS score of <27
6. Current shift worker
7. Resides in a nursing home
8. Unstable medical condition (e.g., unstable angina, end stage renal disease)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation over 12 months using the Beck Scale for Suicidal Ideation (BSSI) | Baseline and at month 1, 2, 3, 6, 9, and 12.
  The BSSI is one of the most commonly used clinician-administered scales to assess presence and severity of suicidality. The total BSS score can range from 0 to 38, with higher values indicating a greater risk of suicide.
Change in perceived loneliness over 12 months using the UCLA Loneliness Scale | Baseline and at month 1, 2, 3, 6, 9, and 12.
  The UCLA Loneliness Scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. The total score ranges from 20 to 80. Higher scores indicate higher loneliness.

SECONDARY OUTCOMES:
Interdaily stability of the rest-activity rhythm | Baseline and at month 1, 2, 3, 6, 9, and 12.
  Measured using 1-week of accelerometry recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Stahl, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh (UPMC), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No